CLINICAL TRIAL: NCT03356652
Title: Electrical Activation Mapping Guided Tailor Made Approach for Cardiac Resynchronization Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Bryan Ping Yen YAN, Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CUHK-MAPCRT-1
Record Dates: First submitted 2017-11-08; First posted 2017-11-29 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure
Keywords: Cardiac resynchronizaton therapy; Electrical activation mapping; Noninvasive; Electrical dyssynchrony
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tailor-made CRT delivery (Experimental): Patient undergoes acute noninvasive electrical dyssynchrony study with various CRT configurations. CRT device is then implanted with optimal configuration.
  Interventions: Procedure: Noninvasive electrical dyssynchrony study

INTERVENTIONS:
Procedure: Noninvasive electrical dyssynchrony study — Ventricular activation maps will be acquired simultaneously with hemodynamic measurements using noninvasive mapping system (ECVUE, Medtronic Inc, USA). A thoracic computed tomographic scan will be acquired with the electrodes attached to the patient. Local ventricular activation times will be defined as the onset of the QRS complex or the pacing spike to the maximal negative slope of each unipolar electrogram.
  Pacing leads will be placed in high right atrium, His-bundle region, right ventricular apex, high septal RV, coronary sinus posterior/lateral branch, coronary sinus anterior branch, lateral and septal region of endocardial LV in order to deliver CRT in 8 different configurations.
  Other Names: Noninvasive electrical activation; Electrical Activation Mapping; Noninvasive mapping system; ECVUE

SUMMARY:
Background

Cardiac Resynchronization Therapy (CRT) is proven to improve survival and heart function of patient with certain electrical conduction abnormality and heart failure. However, in patient with certain electrical conduction abnormality, a good response is observed in less than 40% in patient receiving CRT. Conventionally the surgical approach of CRT is to implant one pacing lead in the right heart and one in the left heart to resynchronize the contraction and the pacing lead in the left heart is usually placed in the posterior or lateral portion of the left heart. However, this single approach may not be optimal, especially for those patients with conduction abnormality known to have poor response to CRT.

Purpose of the clinical investigation

The purpose of the Electrical Activation Guided CRT Study is to study the effectiveness of a tailored made approach to CRT procedure by using a noninvasive globally mapping system studying the electrical conduction under different approaches to delivery CRT. The pacing approach that optimally corrects conduction abnormality will be determined before the actual implantation procedure.

Conduct of the Investigation

This study will include 93 patients with conduction abnormality that known to have a poor response to CRT from Prince of Wales Hospital, Hong Kong.Subjects will be followed up at 3 months and 6 months visit.

DETAILED DESCRIPTION:
The purpose is to prospectively study the feasibility to optimize configuration of CRT delivery for acute correction of electrical dyssynchrony using a noninvasive mapping of global electrical activation.

Study Hypothesis: Tailor-made configuration of CRT delivery is feasible and able to improve responder rate compare to single method of CRT delivery in candidates with known poor response to CRT.

Primary outcome measure: Responder rate of greater than 10% of LV end systolic volume reduction in patients undergoing tailor-made approach of CRT delivery at 6 months. The responder rate is to compare with pre-defined level of 40% for single method of CRT delivery namely biventricular pacing with LV lead in coronary sinus.

Sample Size: The total required sample size is 93 patients with device implanted.

ELIGIBILITY:
Inclusion Criteria:

* Adult (aged 18 or above) of both sexes
* Ischemic or non-ischemic cause of heart failure
* QRS duration > 120 ms, non -LBBB type of conduction disturbance
* NYHA class III or above
* Sinus rhythm
* Informed consent by the patient
* Already received stable dose of guideline directed medical therapy for at least 3 months

Exclusion Criteria:

* LBBB* patients
* Pregnant women
* Participation in another study
* Patient with contraindication to left ventricle catheterization by a retrograde aortic approach (eg mechanical aortic valve, severe aortic stenosis and aortic dissection) *The definitions of LBBB (QRS duration ≥130 ms; QS or rS in lead V1; broad R waves in leads I, aVL, V5, or V6; and absent q waves in leads I, V5, and V6).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2018-03-08 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Responder rate of greater than 10% of LV end systolic volume reduction in patients undergoing tailor-made approach of CRT delivery at 6 months. | 6 months
  Responder rate of greater than 10% of LV end systolic volume reduction measured by echocardiogram comparing baseline and 6 months post implant in patients undergoing tailor-made approach of CRT delivery. Responder rate of greater than 10% of LV end systolic volume reduction measured by echocardiogram comparing baseline and 6 months post implant in patients undergoing tailor-made approach of CRT delivery. The responder rate is to compare with pre-defined level of 40% for single method of CRT delivery namely biventricular pacing with LV lead in coronary sinus.

SECONDARY OUTCOMES:
The acute electrical dyssynchrony indices of different methods of CRT delivery. | during procedure
  The acute electrical dyssynchrony indices of different methods of CRT delivery.
The hemodynamic responses of different methods of CRT delivery. | during procedure
  The hemodynamic responses of different methods of CRT delivery. The hemodynamic response will be maximal dp/dt as measured by pressure wire introduced into the left ventricle during the procedure.
Procedure duration of the optimal CRT delivery method | during procedure
  Procedure duration of the optimal CRT delivery method as determined by the best improvement in electrical dyssynchrony indices.
Implantation success rate of the optimal CRT delivery method | during procedure
  Implantation success rate of the optimal CRT delivery method as determined by the best improvement in electrical dyssynchrony indices.
Cine images (PA, LAO 300, RAO 300) and Chest X ray (PA view) | during procedure
  Cine images (PA, LAO 300, RAO 300) and Chest X ray (PA view)
Peri-operative and 6 months follow-up complications rate: | Peri-operative and 6 months
  1. Thromboembolic event
  2. Dislodgement and migration of pacing leads
  3. Phrenic nerve stimulation
  4. Others
Left ventricular systolic and diastolic volume at baseline and 6 months: | baseline and 6 months
  Echocardiogram parameter of left ventricular systolic and diastolic volume at baseline and 6 months.
Left ventricular ejection fraction at baseline and 6 months: | baseline and 6 months
  Echocardiogram parameter of left ventricular ejection fraction at baseline and 6 months.
Degree of mitral regurgitation at baseline and 6 months: | baseline and 6 months
  Echocardiogram parameter of degree of mitral regurgitation at baseline and 6 months.
Strain imaging at baseline and 6 months: | baseline and 6 months
  Echocardiogram parameter of strain imaging at baseline and 6 months.
NYHA class | baseline and 6 months
  NYHA class at baseline and 6 months.
6 minute hall walk test | baseline and 6 months
  6 minute hall walk test at baseline and 6 months.
Quality of life using Minnesota's questionnaire | baseline and 6 months
  Quality of life using Minnesota's questionnaire at baseline and 6 months.
Electrical parameters including threshold, sensitivity and lead impedance of pacing leads at implant and 6 months follow-up. | during procedure and 6 months
  Electrical parameters including threshold, sensitivity and lead impedance of pacing leads at implant and 6 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan PY YAN, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bristow MR, Saxon LA, Boehmer J, Krueger S, Kass DA, De Marco T, Carson P, DiCarlo L, DeMets D, White BG, DeVries DW, Feldman AM; Comparison of Medical Therapy, Pacing, and Defibrillation in Heart Failure (COMPANION) Investigators. Cardiac-resynchronization therapy with or without an implantable defibrillator in advanced chronic heart failure. N Engl J Med. 2004 May 20;350(21):2140-50. doi: 10.1056/NEJMoa032423. PMID 15152059
- [Background] Cleland JG, Daubert JC, Erdmann E, Freemantle N, Gras D, Kappenberger L, Tavazzi L; Cardiac Resynchronization-Heart Failure (CARE-HF) Study Investigators. The effect of cardiac resynchronization on morbidity and mortality in heart failure. N Engl J Med. 2005 Apr 14;352(15):1539-49. doi: 10.1056/NEJMoa050496. Epub 2005 Mar 7. PMID 15753115
- [Background] Tang AS, Wells GA, Talajic M, Arnold MO, Sheldon R, Connolly S, Hohnloser SH, Nichol G, Birnie DH, Sapp JL, Yee R, Healey JS, Rouleau JL; Resynchronization-Defibrillation for Ambulatory Heart Failure Trial Investigators. Cardiac-resynchronization therapy for mild-to-moderate heart failure. N Engl J Med. 2010 Dec 16;363(25):2385-95. doi: 10.1056/NEJMoa1009540. Epub 2010 Nov 14. PMID 21073365
- [Background] Bradley DJ, Bradley EA, Baughman KL, Berger RD, Calkins H, Goodman SN, Kass DA, Powe NR. Cardiac resynchronization and death from progressive heart failure: a meta-analysis of randomized controlled trials. JAMA. 2003 Feb 12;289(6):730-40. doi: 10.1001/jama.289.6.730. PMID 12585952
- [Background] Cleland JG, Abraham WT, Linde C, Gold MR, Young JB, Claude Daubert J, Sherfesee L, Wells GA, Tang AS. An individual patient meta-analysis of five randomized trials assessing the effects of cardiac resynchronization therapy on morbidity and mortality in patients with symptomatic heart failure. Eur Heart J. 2013 Dec;34(46):3547-56. doi: 10.1093/eurheartj/eht290. Epub 2013 Jul 29. PMID 23900696
- [Background] European Society of Cardiology (ESC); European Heart Rhythm Association (EHRA); Brignole M, Auricchio A, Baron-Esquivias G, Bordachar P, Boriani G, Breithardt OA, Cleland J, Deharo JC, Delgado V, Elliott PM, Gorenek B, Israel CW, Leclercq C, Linde C, Mont L, Padeletti L, Sutton R, Vardas PE. 2013 ESC guidelines on cardiac pacing and cardiac resynchronization therapy: the task force on cardiac pacing and resynchronization therapy of the European Society of Cardiology (ESC). Developed in collaboration with the European Heart Rhythm Association (EHRA). Europace. 2013 Aug;15(8):1070-118. doi: 10.1093/europace/eut206. Epub 2013 Jun 24. No abstract available. PMID 23801827
- [Background] Russo AM, Stainback RF, Bailey SR, Epstein AE, Heidenreich PA, Jessup M, Kapa S, Kremers MS, Lindsay BD, Stevenson LW. ACCF/HRS/AHA/ASE/HFSA/SCAI/SCCT/SCMR 2013 appropriate use criteria for implantable cardioverter-defibrillators and cardiac resynchronization therapy: a report of the American College of Cardiology Foundation appropriate use criteria task force, Heart Rhythm Society, American Heart Association, American Society of Echocardiography, Heart Failure Society of America, Society for Cardiovascular Angiography and Interventions, Society of Cardiovascular Computed Tomography, and Society for Cardiovascular Magnetic Resonance. J Am Coll Cardiol. 2013 Mar 26;61(12):1318-68. doi: 10.1016/j.jacc.2012.12.017. Epub 2013 Mar 1. No abstract available. PMID 23453819
- [Background] Sipahi I, Chou JC, Hyden M, Rowland DY, Simon DI, Fang JC. Effect of QRS morphology on clinical event reduction with cardiac resynchronization therapy: meta-analysis of randomized controlled trials. Am Heart J. 2012 Feb;163(2):260-7.e3. doi: 10.1016/j.ahj.2011.11.014. PMID 22305845
- [Background] Peterson PN, Greiner MA, Qualls LG, Al-Khatib SM, Curtis JP, Fonarow GC, Hammill SC, Heidenreich PA, Hammill BG, Piccini JP, Hernandez AF, Curtis LH, Masoudi FA. QRS duration, bundle-branch block morphology, and outcomes among older patients with heart failure receiving cardiac resynchronization therapy. JAMA. 2013 Aug 14;310(6):617-26. doi: 10.1001/jama.2013.8641. PMID 23942680
- [Background] Eschalier R, Ploux S, Ritter P, Haissaguerre M, Ellenbogen KA, Bordachar P. Nonspecific intraventricular conduction delay: Definitions, prognosis, and implications for cardiac resynchronization therapy. Heart Rhythm. 2015 May;12(5):1071-9. doi: 10.1016/j.hrthm.2015.01.023. Epub 2015 Jan 19. PMID 25614250
- [Background] Nery PB, Ha AC, Keren A, Birnie DH. Cardiac resynchronization therapy in patients with left ventricular systolic dysfunction and right bundle branch block: a systematic review. Heart Rhythm. 2011 Jul;8(7):1083-7. doi: 10.1016/j.hrthm.2011.01.041. Epub 2011 Feb 4. PMID 21300176
- [Background] Byrne MJ, Helm RH, Daya S, Osman NF, Halperin HR, Berger RD, Kass DA, Lardo AC. Diminished left ventricular dyssynchrony and impact of resynchronization in failing hearts with right versus left bundle branch block. J Am Coll Cardiol. 2007 Oct 9;50(15):1484-90. doi: 10.1016/j.jacc.2007.07.011. Epub 2007 Sep 24. PMID 17919569
- [Background] Gold MR, Thebault C, Linde C, Abraham WT, Gerritse B, Ghio S, St John Sutton M, Daubert JC. Effect of QRS duration and morphology on cardiac resynchronization therapy outcomes in mild heart failure: results from the Resynchronization Reverses Remodeling in Systolic Left Ventricular Dysfunction (REVERSE) study. Circulation. 2012 Aug 14;126(7):822-9. doi: 10.1161/CIRCULATIONAHA.112.097709. Epub 2012 Jul 10. PMID 22781424
- [Background] Hara H, Oyenuga OA, Tanaka H, Adelstein EC, Onishi T, McNamara DM, Schwartzman D, Saba S, Gorcsan J 3rd. The relationship of QRS morphology and mechanical dyssynchrony to long-term outcome following cardiac resynchronization therapy. Eur Heart J. 2012 Nov;33(21):2680-91. doi: 10.1093/eurheartj/ehs013. Epub 2012 Feb 19. PMID 22351700
- [Background] Haghjoo M, Bagherzadeh A, Farahani MM, Haghighi ZO, Sadr-Ameli MA. Significance of QRS morphology in determining the prevalence of mechanical dyssynchrony in heart failure patients eligible for cardiac resynchronization: particular focus on patients with right bundle branch block with and without coexistent left-sided conduction defects. Europace. 2008 May;10(5):566-71. doi: 10.1093/europace/eun081. Epub 2008 Apr 3. PMID 18390536
- [Background] Ghosh S, Silva JN, Canham RM, Bowman TM, Zhang J, Rhee EK, Woodard PK, Rudy Y. Electrophysiologic substrate and intraventricular left ventricular dyssynchrony in nonischemic heart failure patients undergoing cardiac resynchronization therapy. Heart Rhythm. 2011 May;8(5):692-9. doi: 10.1016/j.hrthm.2011.01.017. Epub 2011 Jan 11. PMID 21232630
- [Background] Ploux S, Eschalier R, Whinnett ZI, Lumens J, Derval N, Sacher F, Hocini M, Jais P, Dubois R, Ritter P, Haissaguerre M, Wilkoff BL, Francis DP, Bordachar P. Electrical dyssynchrony induced by biventricular pacing: implications for patient selection and therapy improvement. Heart Rhythm. 2015 Apr;12(4):782-91. doi: 10.1016/j.hrthm.2014.12.031. Epub 2014 Dec 26. PMID 25546811
- [Background] Ploux S, Lumens J, Whinnett Z, Montaudon M, Strom M, Ramanathan C, Derval N, Zemmoura A, Denis A, De Guillebon M, Shah A, Hocini M, Jais P, Ritter P, Haissaguerre M, Wilkoff BL, Bordachar P. Noninvasive electrocardiographic mapping to improve patient selection for cardiac resynchronization therapy: beyond QRS duration and left bundle branch block morphology. J Am Coll Cardiol. 2013 Jun 18;61(24):2435-2443. doi: 10.1016/j.jacc.2013.01.093. Epub 2013 Apr 16. PMID 23602768
- [Background] Auricchio A, Fantoni C, Regoli F, Carbucicchio C, Goette A, Geller C, Kloss M, Klein H. Characterization of left ventricular activation in patients with heart failure and left bundle-branch block. Circulation. 2004 Mar 9;109(9):1133-9. doi: 10.1161/01.CIR.0000118502.91105.F6. Epub 2004 Mar 1. PMID 14993135
- [Background] Auricchio A, Lumens J, Prinzen FW. Does cardiac resynchronization therapy benefit patients with right bundle branch block: cardiac resynchronization therapy has a role in patients with right bundle branch block. Circ Arrhythm Electrophysiol. 2014 Jun;7(3):532-42. doi: 10.1161/CIRCEP.113.000628. No abstract available. PMID 24951571
- [Background] Varma N, Jia P, Rudy Y. Electrocardiographic imaging of patients with heart failure with left bundle branch block and response to cardiac resynchronization therapy. J Electrocardiol. 2007 Nov-Dec;40(6 Suppl):S174-8. doi: 10.1016/j.jelectrocard.2007.06.017. PMID 17993318
- [Background] Lund LH, Jurga J, Edner M, Benson L, Dahlstrom U, Linde C, Alehagen U. Prevalence, correlates, and prognostic significance of QRS prolongation in heart failure with reduced and preserved ejection fraction. Eur Heart J. 2013 Feb;34(7):529-39. doi: 10.1093/eurheartj/ehs305. Epub 2012 Oct 4. PMID 23041499
- [Background] Khan FZ, Virdee MS, Palmer CR, Pugh PJ, O'Halloran D, Elsik M, Read PA, Begley D, Fynn SP, Dutka DP. Targeted left ventricular lead placement to guide cardiac resynchronization therapy: the TARGET study: a randomized, controlled trial. J Am Coll Cardiol. 2012 Apr 24;59(17):1509-18. doi: 10.1016/j.jacc.2011.12.030. Epub 2012 Mar 7. PMID 22405632
- [Background] Gold MR, Birgersdotter-Green U, Singh JP, Ellenbogen KA, Yu Y, Meyer TE, Seth M, Tchou PJ. The relationship between ventricular electrical delay and left ventricular remodelling with cardiac resynchronization therapy. Eur Heart J. 2011 Oct;32(20):2516-24. doi: 10.1093/eurheartj/ehr329. Epub 2011 Aug 29. PMID 21875862
- [Background] Lustgarten DL, Crespo EM, Arkhipova-Jenkins I, Lobel R, Winget J, Koehler J, Liberman E, Sheldon T. His-bundle pacing versus biventricular pacing in cardiac resynchronization therapy patients: A crossover design comparison. Heart Rhythm. 2015 Jul;12(7):1548-57. doi: 10.1016/j.hrthm.2015.03.048. Epub 2015 Mar 28. PMID 25828601
- [Background] Anselme F, Bordachar P, Pasquie JL, Klug D, Leclercq C, Milhem A, Alonso C, Deharo JC, Gras D, Probst V, Piot O, Savoure A. Safety, feasibility, and outcome results of cardiac resynchronization with triple-site ventricular stimulation compared to conventional cardiac resynchronization. Heart Rhythm. 2016 Jan;13(1):183-9. doi: 10.1016/j.hrthm.2015.08.036. Epub 2015 Sep 26. PMID 26325531
- [Background] Lenarczyk R, Kowalski O, Sredniawa B, Pruszkowska-Skrzep P, Mazurek M, Jedrzejczyk-Patej E, Wozniak A, Pluta S, Glowacki J, Kalarus Z. Implantation feasibility, procedure-related adverse events and lead performance during 1-year follow-up in patients undergoing triple-site cardiac resynchronization therapy: a substudy of TRUST CRT randomized trial. J Cardiovasc Electrophysiol. 2012 Nov;23(11):1228-36. doi: 10.1111/j.1540-8167.2012.02375.x. Epub 2012 May 31. PMID 22651239
- [Background] Bordachar P, Alonso C, Anselme F, Boveda S, Defaye P, Garrigue S, Gras D, Klug D, Piot O, Sadoul N, Leclercq C. Addition of a second LV pacing site in CRT nonresponders rationale and design of the multicenter randomized V(3) trial. J Card Fail. 2010 Sep;16(9):709-13. doi: 10.1016/j.cardfail.2010.04.010. Epub 2010 Jun 8. PMID 20797593
- [Background] Morgan JM, Biffi M, Geller L, Leclercq C, Ruffa F, Tung S, Defaye P, Yang Z, Gerritse B, van Ginneken M, Yee R, Jais P; ALSYNC Investigators. ALternate Site Cardiac ResYNChronization (ALSYNC): a prospective and multicentre study of left ventricular endocardial pacing for cardiac resynchronization therapy. Eur Heart J. 2016 Jul 14;37(27):2118-27. doi: 10.1093/eurheartj/ehv723. Epub 2016 Jan 18. PMID 26787437
- [Background] Fang F, Zhang Q, Chan JY, Razali O, Azlan H, Chan HC, Sanderson JE, Xie JM, Yu CM. Early pacing-induced systolic dyssynchrony is a strong predictor of left ventricular adverse remodeling: analysis from the Pacing to Avoid Cardiac Enlargement (PACE) trial. Int J Cardiol. 2013 Sep 30;168(2):723-8. doi: 10.1016/j.ijcard.2012.08.005. Epub 2012 Sep 1. PMID 22944596
- [Background] Zhang Q, van Bommel RJ, Chan YS, Delgado V, Liang Y, Schalij MJ, Bax JJ, Fang F, Wai-Kwok Yip G, Yu CM. Diverse patterns of longitudinal and radial dyssynchrony in patients with advanced systolic heart failure. Heart. 2011 Apr;97(7):574-8. doi: 10.1136/hrt.2010.198572. Epub 2011 Jan 30. PMID 21282133
- [Background] Fang F, Chan JY, Yip GW, Xie JM, Zhang Q, Fung JW, Lam YY, Yu CM. Prevalence and determinants of left ventricular systolic dyssynchrony in patients with normal ejection fraction received right ventricular apical pacing: a real-time three-dimensional echocardiographic study. Eur J Echocardiogr. 2010 Mar;11(2):109-18. doi: 10.1093/ejechocard/jep171. Epub 2009 Nov 20. PMID 19933290
- [Background] Zhang Q, van Bommel RJ, Fung JW, Chan JY, Bleeker GB, Ypenburg C, Yip G, Liang YJ, Schalij MJ, Bax JJ, Yu CM. Tissue Doppler velocity is superior to strain imaging in predicting long-term cardiovascular events after cardiac resynchronisation therapy. Heart. 2009 Jul;95(13):1085-90. doi: 10.1136/hrt.2008.161653. Epub 2009 Apr 9. PMID 19363024
- [Background] Zhang Q, Fang F, Yip GW, Chan JY, Shang Q, Fung JW, Chan AK, Liang YJ, Yu CM. Difference in prevalence and pattern of mechanical dyssynchrony in left bundle branch block occurring in right ventricular apical pacing versus systolic heart failure. Am Heart J. 2008 Nov;156(5):989-95. doi: 10.1016/j.ahj.2008.06.027. Epub 2008 Sep 11. PMID 19061717
- [Background] Fung JW, Lam YY, Zhang Q, Yip GW, Chan WW, Chan GC, Chan JY, Yu CM. Effect of left ventricular lead concordance to the delayed contraction segment on echocardiographic and clinical outcomes after cardiac resynchronization therapy. J Cardiovasc Electrophysiol. 2009 May;20(5):530-5. doi: 10.1111/j.1540-8167.2008.01364.x. Epub 2008 Nov 21. PMID 19054250
- [Background] Zhang Y, Yip GW, Chan AK, Wang M, Lam WW, Fung JW, Chan JY, Sanderson JE, Yu CM. Left ventricular systolic dyssynchrony is a predictor of cardiac remodeling after myocardial infarction. Am Heart J. 2008 Dec;156(6):1124-32. doi: 10.1016/j.ahj.2008.07.019. Epub 2008 Oct 26. PMID 19033008
- [Background] Zhang Q, Fung JW, Chan JY, Yip G, Lam YY, Liang YJ, Yu CM. Difference in long-term clinical outcome after cardiac resynchronisation therapy between ischaemic and non-ischaemic aetiologies of heart failure. Heart. 2009 Feb;95(2):113-8. doi: 10.1136/hrt.2008.145698. Epub 2008 Jul 24. PMID 18653570
- [Background] Zhang Q, Fung JW, Yip GW, Chan JY, Lee AP, Lam YY, Wu LW, Wu EB, Yu CM. Improvement of left ventricular myocardial short-axis, but not long-axis function or torsion after cardiac resynchronisation therapy: an assessment by two-dimensional speckle tracking. Heart. 2008 Nov;94(11):1464-71. doi: 10.1136/hrt.2007.127498. Epub 2008 Jan 15. PMID 18198202
- [Background] Van de Veire NR, Yu CM, Ajmone-Marsan N, Bleeker GB, Ypenburg C, De Sutter J, Zhang Q, Fung JW, Chan JY, Holman ER, van der Wall EE, Schalij MJ, Bax JJ. Triplane tissue Doppler imaging: a novel three-dimensional imaging modality that predicts reverse left ventricular remodelling after cardiac resynchronisation therapy. Heart. 2008 Mar;94(3):e9. doi: 10.1136/hrt.2007.122564. Epub 2007 Nov 5. PMID 17984218
- [Background] Yu CM, Gorcsan J 3rd, Bleeker GB, Zhang Q, Schalij MJ, Suffoletto MS, Fung JW, Schwartzman D, Chan YS, Tanabe M, Bax JJ. Usefulness of tissue Doppler velocity and strain dyssynchrony for predicting left ventricular reverse remodeling response after cardiac resynchronization therapy. Am J Cardiol. 2007 Oct 15;100(8):1263-70. doi: 10.1016/j.amjcard.2007.05.060. Epub 2007 Aug 20. PMID 17920368
- [Background] Fung JW, Chan JY, Yip GW, Chan HC, Chan WW, Zhang Q, Yu CM. Effect of left ventricular endocardial activation pattern on echocardiographic and clinical response to cardiac resynchronization therapy. Heart. 2007 Apr;93(4):432-7. doi: 10.1136/hrt.2007.115295. Epub 2007 Jan 19. PMID 17237127
- [Background] Yu CM, Chan YS, Zhang Q, Yip GW, Chan CK, Kum LC, Wu L, Lee AP, Lam YY, Fung JW. Benefits of cardiac resynchronization therapy for heart failure patients with narrow QRS complexes and coexisting systolic asynchrony by echocardiography. J Am Coll Cardiol. 2006 Dec 5;48(11):2251-7. doi: 10.1016/j.jacc.2006.07.054. PMID 17161255
- [Background] Yu CM, Zhang Q, Yip GW, Chan YS, Lee PW, Wu LW, Lam YY, Kum LC, Chan HC, Chan S, Fung JW. Are left ventricular diastolic function and diastolic asynchrony important determinants of response to cardiac resynchronization therapy? Am J Cardiol. 2006 Oct 15;98(8):1083-7. doi: 10.1016/j.amjcard.2006.05.028. Epub 2006 Aug 30. PMID 17027576
- [Background] Fung JW, Zhang Q, Yip GW, Chan JY, Chan HC, Yu CM. Effect of cardiac resynchronization therapy in patients with moderate left ventricular systolic dysfunction and wide QRS complex: a prospective study. J Cardiovasc Electrophysiol. 2006 Dec;17(12):1288-92. doi: 10.1111/j.1540-8167.2006.00612.x. Epub 2006 Sep 20. PMID 16987381
- [Background] Yu CM, Zhang Q, Fung JW, Chan HC, Chan YS, Yip GW, Kong SL, Lin H, Zhang Y, Sanderson JE. A novel tool to assess systolic asynchrony and identify responders of cardiac resynchronization therapy by tissue synchronization imaging. J Am Coll Cardiol. 2005 Mar 1;45(5):677-84. doi: 10.1016/j.jacc.2004.12.003. PMID 15734610
- [Background] Zhang Q, Yu CM, Fung JW, Zhang Y, Chan YS, Chan HC, Yip GW, Sanderson JE. Assessment of the effect of cardiac resynchronization therapy on intraventricular mechanical synchronicity by regional volumetric changes. Am J Cardiol. 2005 Jan 1;95(1):126-9. doi: 10.1016/j.amjcard.2004.08.078. PMID 15619410
- [Background] Chung ES, Leon AR, Tavazzi L, Sun JP, Nihoyannopoulos P, Merlino J, Abraham WT, Ghio S, Leclercq C, Bax JJ, Yu CM, Gorcsan J 3rd, St John Sutton M, De Sutter J, Murillo J. Results of the Predictors of Response to CRT (PROSPECT) trial. Circulation. 2008 May 20;117(20):2608-16. doi: 10.1161/CIRCULATIONAHA.107.743120. Epub 2008 May 5. PMID 18458170

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT03356652/Prot_SAP_000.pdf